CLINICAL TRIAL: NCT05814393
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel, Phase Ⅲ Study to Evaluate the Efficacy and Safety of JW0201 Added on in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control With C2202 and C2203
Brief Title: To Evaluate the Efficacy and Safety of JW0201 Added on in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JW22301
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JW0201+C2202+C2203 (Experimental): Treatment period for 24 weeks (After the treatment period, take JW0201+C2202+C2203 for 28 weeks)
  Interventions: Drug: Treatment Period(JW0201); Drug: Extension Period(JW0201)
- C2202+C2203 (Placebo Comparator): Treatment period for 24 weeks (After the treatment period, take JW0201+C2202+C2203 for 28 weeks)
  Interventions: Drug: Treatment Period(Placebo); Drug: Extension Period(JW0201)

INTERVENTIONS:
Drug: Treatment Period(JW0201) — JW0201: 200mg/day For 24 weeks(PO, BID) C2022: ≥1,000 mg/day for 24 Weeks(PO, BID) C2203: 25 mg/day for 24 Weeks(PO, BID)
  Other Names: JW0201+C2022+C2203
  Arms: JW0201+C2202+C2203
Drug: Treatment Period(Placebo) — C2022: ≥1,000 mg/day for 24 Weeks(PO, BID) C2203: 25 mg/day for 24 Weeks(PO, BID)
  Other Names: C2022+C2203
  Arms: C2202+C2203
Drug: Extension Period(JW0201) — JW0201: 200mg/day For 28 weeks(PO, BID) C2022: ≥1,000 mg/day for 28 Weeks(PO, BID) C2203: 25 mg/day for 28 Weeks(PO, BID)
  Other Names: JW0201+C2022+C2203

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, parallel, phase Ⅲ study to evaluate the efficacy and safety of JW0201 added on in patients with type 2 diabetes mellitus who have inadequate glycemic control with C2202 and C2203

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled, parallel, phase Ⅲ study

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* The subject not meet the specified HbA1c and FPG

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
HbA1c (24 Weeks) lowering effect | 24 Weeks
  change in HbA1c

SECONDARY OUTCOMES:
HbA1c lowering effect | 6, 12, 18, 32, 40, 52 Weeks
  change in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-Young Park, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea